CLINICAL TRIAL: NCT06133023
Title: WONDER-02: Plastic Stent vs. Lumen-apposing Metal Stent for Endoscopic Ultrasound-guided Drainage of Pancreatic Pseudocysts-a Multicentre Randomised Non-inferiority Trial
Brief Title: WONDER-02 Trial: Plastic Stent vs. Lumen-apposing Metal Stent for Pancreatic Pseudocysts
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tokyo University (Other)
Responsible Party: Principal Investigator, Yousuke Nakai, Associate professor, Department of Endoscopy and Endoscopic Surgery, The University of Tokyo Hospital, Tokyo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023002P
Record Dates: First submitted 2023-10-29; First posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Pancreatic Fluid Collection; Pancreatitis; Pancreatic Pseudocyst
Keywords: Endosonography; Drainage; Stents; Pancreatic Pseudocyst
MeSH Terms: conditions — Pancreatitis; Pancreatic Pseudocyst

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plastic stent group (Experimental): In the plastic stent group, two (at least one) 7-Fr double pigtail stents will be placed. Following EUS-guided puncture of a pseudocyst, a guidewire will be coiled within the lesion, and another guidewire will be inserted alongside the prepositioned guidewire. The puncture tract will be dilated if needed.
  Interventions: Procedure: Plastic stent
- LAMS group (Active Comparator): In the LAMS group, a LAMS with electrocautery enhanced delivery will be placed (Hot AXIOS; Boston Scientific Japan, Tokyo, Japan). A guidewire or dilator will be used if needed.
  Interventions: Procedure: LAMS

INTERVENTIONS:
Procedure: Plastic stent — EUS-guided drainage will be conducted under endosonographic and fluoroscopic guidance within 72 hours of the randomisation. A linear echoendoscope will be advanced to the stomach or duodenum with moderate sedation, and the targeted pseudocyst will be visualised and punctured under endosonographic guidance. In cases with an insufficient improvement in inflammatory indicators (i.e., body temperature, white blood cell count, and C-reactive protein), the investigators will perform additional interventions including the addition of or replacement with a plastic stent or LAMS and/or percutaneous drainage if needed.
  In the plastic stent group, two (at least one) 7-Fr double pigtail stents will be placed. Following EUS-guided puncture of a pseudocyst, a guidewire will be coiled within the lesion, and another guidewire will be inserted alongside the prepositioned guidewire. The puncture tract will be dilated if needed.
  Arms: Plastic stent group
Procedure: LAMS — EUS-guided drainage will be conducted under endosonographic and fluoroscopic guidance within 72 hours of the randomisation. A linear echoendoscope will be advanced to the stomach or duodenum with moderate sedation, and the targeted pseudocyst will be visualised and punctured under endosonographic guidance. In cases with an insufficient improvement in inflammatory indicators (i.e., body temperature, white blood cell count, and C-reactive protein), the investigators will perform additional interventions including the addition of or replacement with a plastic stent or LAMS and/or percutaneous drainage if needed.
  In the LAMS group, a LAMS with electrocautery enhanced delivery will be placed (Hot AXIOS; Boston Scientific Japan, Tokyo, Japan). A guidewire or dilator will be used if needed.
  Arms: LAMS group

SUMMARY:
Endoscopic ultrasound (EUS)-guided transluminal drainage has become a first-line treatment modality for symptomatic pancreatic pseudocysts. Despite the increasing popularity of lumen-apposing metal stents (LAMSs), the use of a LAMS is limited by its high costs and specific adverse events compared to plastic stent placement. To date, there has been a paucity of data on the appropriate stent type in this setting. This trial aims to assess the non-inferiority of plastic stents to a LAMS for the initial EUS-guided drainage of pseudocysts.

DETAILED DESCRIPTION:
Pancreatic fluid collections (PFCs) develop as local complications of acute pancreatitis after four weeks of the disease onset. Pancreatic pseudocysts are a type of PFC, which is characterised by encapsulated non-necrotic contents. Pseudocysts occasionally become symptomatic (e.g., infection, GI symptoms), and given the high morbidity and mortality, it is mandatory to manage symptomatic pseudocysts appropriately to improve clinical outcomes of patients with acute pancreatitis overall. EUS-guided transluminal drainage has become a first-choice treatment option for symptomatic PFCs. In the setting of EUS-guided treatment of walled-off necrosis (WON, the other type of PFC), the potential benefits of LAMSs have been reported. Compared to plastic stents, LAMSs can serve as a transluminal port and thereby, facilitate the treatment of WON that often requires a long treatment duration with repeated interventions including direct endoscopic necrosectomy. With the increasing popularity and availability of LAMSs in interventional EUS overall, several retrospective studies have reported the feasibility of LAMS use for EUS-guided drainage of pancreatic pseudocysts.

While a LAMS may enhance the drainage efficiency of pseudocysts due to its large calibre, the benefits of this stent may be mitigated in pseudocysts that, by definition, contain non-necrotic liquid contents and can be managed without necrosectomy. Indeed, several retrospective comparative studies failed to demonstrate the superiority of plastic stents to a LAMS. In addition, the use of a LAMS has been limited by higher costs compared to plastic stents and potential specific adverse events (e.g., bleeding, buried stent). Studies suggest that a prolonged duration of LAMS placement (approximately ≥ 4 weeks) may predispose the patients to an elevated risk of adverse events associated with LAMSs. Therefore, patients requiring long-term drainage (e.g., cases with disconnected pancreatic duct syndrome) should be subjected to a reintervention in which a LAMS is replaced by a plastic stent. However, the technical success rate of the replacement has not been high. Given these lines of evidence, the investigators hypothesised that plastic stents might be non-inferior to a LAMS in terms of the potential of resolving a pseudocyst and associated symptoms.

To test the hypothesis, the investigators have planned a multicentre randomised controlled trial (RCT) to examine the non-inferiority of plastic stents to a LAMS as the initial stent for EUS-guided drainage of pancreatic pseudocysts in terms of the achievement of clinical treatment success (the resolution of a pseudocyst). Given the lower costs of plastic stents compared to a LAMS, the results would help not only establish a new treatment paradigm for pancreatic pseudocysts but also improve the cost-effectiveness of the resource-intensive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pancreatic pseudocyst(s) defined by the revised Atlanta classification
* The longest diameter of a targeted pseudocyst ≥ 5 cm
* Patients requiring drainage for symptoms associated with a pseudocyst (e.g., infection, gastrointestinal symptoms including abdominal pain, or jaundice)
* Patients aged 18 years or older
* Written informed consent obtained from patients or their representatives

Exclusion Criteria:

* A pseudocyst that is inaccessible via the EUS-guided approach
* A plastic or lumen-apposing metal stent in situ
* Coagulopathy (e.g., platelet count < 50,000/mm3 or prothrombin time international normalised ratio [PT-INR] >1.5)
* Users of antithrombotic agents that cannot be discontinued according to the Japan Gastroenterological Endoscopy Society [JGES] guidelines
* Patients who do not tolerate endoscopic procedures
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2033-09 (Estimated)

PRIMARY OUTCOMES:
Clinical success within 180 days of randomisation | Six months
  Clinical success is defined as 1) a decrease in the size of a targeted pancreatic pseudocyst to 2 cm or less and 2) an improvement of at least two out of the following inflammatory indicators: body temperature, white blood cell count, and C-reactive protein.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events | Five years
  The adverse events are defined and graded by the ASGE lexicon guideline.
Mortality | Five years
  Mortality from any cause
Technical success of the initial EUS-guided drainage | One day
  Technical success is defined as the successful placement of any stent in the targeted pseudocyst during the initial EUS-guided drainage.
Time to clinical success | Six months
  Time from randomization to clinical success
Incidence of biliary stricture | Five years
  Biliary stricture due to a pseudocyst
Incidence of gastrointestinal stricture | Five years
  Gastrointestinal obstruction due to a pseudocyst
Time requiring endoscopic drainage | Six months
  Time requiring endoscopic drainage for a pseudocyst
Time requiring percutaneous drainage | Six months
  Time requiring percutaneous drainage for a pseudocyst
Number of interventions | Six months
  Total number of interventions needed for the treatment of a pseudocyst
Time of interventions | Six months
  Total procedure time needed for the treatment of a pseudocyst
Length of the index hospitalisation | Six months
  Total days of the index hospitalisation
Length of ICU stay during the index hospitalisation | Six months
  Total ICU stay of the index hospitalisation
Duration of antibiotics administration | Six months
  Total administration days of antibiotics
Costs of interventions | Six months
  Total costs of treatment interventions
Costs of the index hospitalisation | Six months
  Total costs of the index hospitalisation
Incidence of pseudocyst recurrence | Five years
  Incidence of pseudocyst recurrence after clinical success
Time to recurrence of pancreatic pseudocyst | Five years
  Time from clinical success to recurrence of pancreatic pseudocyst
Treatment duration of recurrent pancreatic pseudocyst | Five years
  Total treatment days for recurrent pancreatic pseudocyst
New onset of pancreatic pseudocyst | Five years
  Incidence of new-onset pancreatic pseudocyst
Treatment duration of new onset pancreatic pseudocyst | Five years
  Total treatment days for new-onset pancreatic pseudocyst
Incidence of new onset diabetes | Five years
  Incidence of new-onset diabetes mellitus
The presence of medications for pancreatic exocrine insufficiency | Five years
  The start of medications for pancreatic exocrine insufficiency and the date
The presence of sarcopenia | Five years
  The presence of sarcopenia and the date of diagnosis
Change in volume of pancreas | Five years
  Change in volume of pancreas. Volume is evaluated by contrast-enhanced Computed Tomography (CT) using SYNAPSE VINCENT (FUJIFILM).
Success rate of surgical procedures | Six months
  Success rate of surgeries associated with pancreatic pseudocyst
Operation time of surgical procedures | Six months
  Total operation times
Incidence of new onset clinical symptoms of pancreatic exocrine insufficiency | Five years
  New-onset clinical symptoms associated with pancreatic exocrine insufficiency, such as steatorrhea , constipation, diarrhea, maldigestion, flatulence, and tenesmus
Incidence of new pancreatic cancer | Five years
  New-onset pancreatic cancer

CONTACTS AND LOCATIONS:
Overall Officials: Yousuke Nakai, Principal Investigator — Department of Endoscopy and Endoscopic Surgery, Graduate School of Medicine, The University of Tokyo
Locations (26):
- Japan (26):
  - Department of Gastroenterology, Aichi Medical University, Aichi
  - Department of Gastroenterology, The University of Tokyo Hospital, Bunkyō-Ku, Tokyo
  - Department of Gastroenterology, Graduate School of Medicine, Juntendo University, Bunkyō-Ku, Tokyo
  - Department of Gastroenterology, Graduate School of Medicine, Chiba University, Chiba
  - Department of Medicine and Bioregulatory Science, Graduate School of Medical Sciences, Kyushu University, Fukuoka
  - Department of Gastroenterology, Gifu Municipal Hospital, Gifu
  - Department of Gastroenterology, Gifu Prefectural General Medical Center, Gifu
  - First Department of Internal Medicine, Gifu University Hospital, Gifu
  - Division of Hepatobiliary and Pancreatic Diseases, Department of Gastroenterology, Hyogo Medical University, Hyōgo
  - Department of Gastroenterology and Neurology, Faculty of Medicine, Kagawa University, Kagawa
  - Digestive and Lifestyle Diseases, Kagoshima University Graduate School of Medical and Dental Sciences, Kagoshima
  - Department of Gastroenterology, Kameda Medical Center, Kamogawa
  - Department of Gastroenterology, St. Marianna University School of Medicine, Kanagawa
  - Department of Gastroenterological Endoscopy, Kanazawa Medical University, Kanazawa
  - Department of Gastroenterology and Hepatology, Saitama Medical Center, Saitama Medical University, Kawagoe
  - Department of Gastroenterology, Teikyo University Mizonokuchi Hospital, Kawasaki
  - Division of Gastroenterology, Department of Internal Medicine, Kobe University Graduate School of Medicine, Kobe
  - Department of Gastroenterology and Hepatology, Mie University Hospital, Mie
  - Department of Gastroenterology and Hepatology, Okayama University Hospital, Okayama
  - 2nd Department of Internal Medicine, Osaka Medical and Pharmaceutical University, Osaka
  - Department of Gastroenterology and Hepatology, Kindai University Faculty of Medicine, Ōsaka
  - Department of Gastroenterology and Hepatology, Hokkaido University Hospital, Sapporo
  - Division of Gastroenterology and Hepatology, Department of Medicine, Nihon University School of Medicine, Tokyo
  - Third Department of Internal Medicine, University of Toyama, Toyama
  - Department of Gastroenterology, Wakayama Medical University School of Medicine, Wakayama
  - Department of Gastroenterology, Yamanashi Prefectural Central Hospital, Yamanashi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Derived] Saito T, Takenaka M, Kuwatani M, Doi S, Ohyama H, Fujisawa T, Masuda A, Iwashita T, Shiomi H, Hayashi N, Iwata K, Maruta A, Mukai T, Matsubara S, Hamada T, Inoue T, Matsumoto K, Hirose S, Fujimori N, Kashiwabara K, Kamada H, Hashimoto S, Shiratori T, Yamada R, Kogure H, Nakahara K, Ogura T, Kitano M, Yasuda I, Isayama H, Nakai Y; WONDERFUL study group in Japan and collaborators. WONDER-02: plastic stent vs. lumen-apposing metal stent for endoscopic ultrasound-guided drainage of pancreatic pseudocysts-study protocol for a multicentre randomised non-inferiority trial. Trials. 2024 Aug 24;25(1):559. doi: 10.1186/s13063-024-08373-6. PMID 39182137